CLINICAL TRIAL: NCT07293715
Title: Permissive Versus Strict Intrapartum Glucose Management in Type 1 Diabetes (PRISM-T1D)
Acronym: PRISM-T1D
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kartik K Venkatesh, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY 20252532
Record Dates: First submitted 2025-12-02; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy, High Risk; Type 1 Diabetes
Keywords: Pregnancy; Continuous Glucose Monitor; Type 1 Diabetes; Automated insulin delivery; Hybrid closed loop; Insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention group (Experimental): permissive blood sugar control (70-140 mg/dL)
  Interventions: Drug: Insulin; Device: DEXCOM Continuous Glucose Monitor
- Standard of care (Other): strict blood sugar control (70-110 mg/dL)
  Interventions: Drug: Insulin; Device: DEXCOM Continuous Glucose Monitor

INTERVENTIONS:
Drug: Insulin — Participants will be randomized in a 1:1 fashion to one of two intrapartum glycemic control options: permissive (70-140 mg/dL) or strict (70-110 mg/dL). Participants and clinicians will be unblinded. Once randomized, an order set will be entered into the EMR that will alert pharmacy and nursing colleagues to the appropriate intrapartum glycemic control protocol.
Device: DEXCOM Continuous Glucose Monitor — Patients will be asked to wear an optional Continuous Glucose Monitor (CGM) to utilize during labor for research purposes. The CGM will be removed prior to hospital discharge and data will be extracted by trained research personnel. All participants already utilize a CGM device as part of standard of care as part of Hybrid Closed Loop (HCL) therapy. No clinical decisions will be made based upon data from the research CGM device. This data will not be extracted until after hospital discharge.

SUMMARY:
PRISM-TID is a single center non-inferiority randomized controlled trial of permissive intrapartum glucose management (intervention) versus strict intrapartum glucose management (standard of care) among pregnant individuals with type 1 diabetes (T1D) using hybrid closed loop therapy (HCL) who are admitted for labor management. Participants will be randomized in a 1:1 fashion to one of two intrapartum glycemic control options: permissive (70-140 mg/dL) or strict (70-110 mg/dL). The primary aim of this trial it to demonstrate that permissive intrapartum glucose management is not associated with an increased risk of neonatal dysglycemia compared with strict intrapartum glucose management.

DETAILED DESCRIPTION:
Type 1 Diabetes (T1D) affects approximately 0.5% of pregnancies in the US. Infants born to individuals with T1D are at increased risk of adverse pregnancy outcomes due to lack of glycemic control. Individuals with T1D are increasingly using hybrid closed loop therapy (HCL) for insulin delivery to achieve glycemic control. Current data highlight that less permissive intrapartum (while in labor) glycemic control is not associated with a increased risk of adverse pregnancy outcomes, including neonatal hypoglycemia and NICU admission. However, such data about permissive versus strict intrapartum glucose management has primarily been from pregnant individuals with type 2 diabetes or gestational diabetes who did not use HCL based insulin therapy. Pregnant individuals with diabetes who use HCL with continuous glucose monitoring and closed loop insulin delivery represent a unique population, and data from this population are needed to inform intrapartum obstetric management. The investigators hypothesize that permissive intrapartum glucose management using continuous glucose monitoring (70-140 mg/dL) will not be associated with neonatal dysglycemia measured as first mean neonatal glucose value within the first two hours of life compared with strict intrapartum glucose management or the current standard of care (70-110 mg/dL). The investigators will conduct a single center non-inferiority randomized controlled trial of permissive intrapartum glucose management (intervention) versus strict intrapartum glucose management (standard of care) among pregnant individuals with T1D using HCL who are admitted for labor management. The primary aim of this trial it to demonstrate that permissive intrapartum glucose management is not associated with an increased risk of neonatal dysglycemia (first neonatal blood glucose measured within 2 hours of life) compared with strict intrapartum glucose management. The investigators will secondarily examine the association between permissive versus strict intrapartum glucose with adverse neonatal outcomes, including neonatal hypoglycemia, neonatal hyperbilirubinemia, and NICU admission, patient satisfaction, and continuous glucose monitor (CGM) metrics.

ELIGIBILITY:
Inclusion Criteria

* Pregnant individuals
* ≥ 18 years old
* Type 1 diabetes utilizing Hybrid Closed Loop (HCL) therapy
* Intention for vaginal delivery and admitted to Labor and Delivery
* Singleton, non-anomalous fetus
* Gestational age greater than or equal to 35 weeks gestation.
* Cervical dilation is less than 6 cm.
* Delivering at the study institution

Exclusion criteria:

* Scheduled cesarean delivery
* Cervical dilation ≥ 6 cm on presentation to L&D
* Receipt of antenatal corticosteroids within 7 days of randomization
* Fetal demise
* Major fetal anomaly (attached)
* Multiple gestation
* Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is restricted to pregnant individuals.
Enrollment: 44 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Mean of first neonatal blood glucose (continuous, mean with standard deviation) | From birth to 2 hours after birth
  The first heel stick neonatal blood glucose (mg/dL) will be obtained within the first two hours of life utilizing a hospital-grade glucometer. This will be recorded in the electronic medical record and abstracted at study conclusion. The mean of these will be utilized as the primary outcome. A heel stick neonatal blood glucose in the first two hours of life is current standard of care for all infants of diabetic individuals.

SECONDARY OUTCOMES:
Neonatal C-peptide (continuous, mean with standard deviation) | At birth
  Umbilical cord C-peptide levels will be analyzed from cord blood collected at the time of delivery.
Neonatal hypoglycemia | At birth, up to 24 hours
  Neonatal hypoglycemia: blood glucose < 40mg/dl in birth to 4 hours of life, < 45mg/dl in 4-24 hours of life, and < 50mg/dl after 24 hours of life, or need for oral or IV glucose therapy.
Neonatal hyperbilirubinemia | Within the first 48 hours after birth
  Neonatal jaundice requiring phototherapy
NICU admission | Within the first 48 hours after birth
  Admitted to NICU during delivery admission
Birth experience satisfaction per Birth Satisfaction Survey-Revised (BSS-R) (continuous, mean with standard deviation) | Day 1 through study completion (at hospital discharge), up to 4 weeks
  The Birth Satisfaction Survey-Revised (BSS-R) is a validated patient satisfaction survey describing L&D birthing experiences. This survey will be administered at any time during their postpartum admission. This measure will be analyzed as a continuous mean score.
Maternal IV insulin maximum dose and duration | Day 1 through study completion, up to 4 weeks
  Maternal IV insulin maximum IV insulin dose (units) and duration (hours) will be measured as continuous variables (mean and SD).
Maternal Hypoglycemia | Day 1 through study completion, up to 4 weeks
  Maternal blood glucose less than 70 mg/dL, as measured by capillary blood glucose via hospital-grade glucometer.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Brewton, MD, Principal Investigator — Ohio State University; Kartik K Venkatesh, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No